CLINICAL TRIAL: NCT00943241
Title: Screening for Breast Cancer in Patients Undergoing Myocardial Perfusion Imaging
Brief Title: Screening in Myocardial Perfusion Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Gamma Medica-Ideas (Industry)
Responsible Party: Principal Investigator, Deborah Rhodes, Assistant Professor of Medicine, Mayo Clinic
Other Study IDs: 08-001046
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Breast; Breast Cancer; MBI; Molecular Breast Imaging; Molecular Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To expand the understanding of the uptake and distribution of Tc-99m sestamibi in the breast in a normal female population undergoing myocardial perfusion imaging using Molecular Breast Imaging (MBI).

DETAILED DESCRIPTION:
You are being asked to take part in this research study because you have been scheduled to have a scan of your heart. The radioactive dye used to image your heart is also taken up by many types of breast cancer. The investigators have developed a new method for detecting breast cancer, called Molecular Breast Imaging that uses this dye.

The purpose of this study is to see how well this new method works in normal subjects with no known breast cancer and to see if we can detect breast cancer at an earlier stage than mammography. As you read this form describing the study, ask any questions you have. Take your time to decide. Feel free to discuss the study with your family, friends, and healthcare provider before you decide. You may stop participating at any time during the study. You may decide not to participate. If so, none of your current benefits or normal health care will be affected in any way. When you feel comfortable that all your questions have been answered, and you wish to take part in this study, sign this form in order to begin your participation. Your signature means you have been told about the study and what the risks are. Your signature on this form also means that you want to take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* They have had a mammogram at Mayo Clinic Rochester within the last 12 months
* Undergoing myocardial perfusion imaging

Exclusion Criteria:

* They are unable to understand and sign the consent form
* They are physically unable to sit upright and still for 20 minutes
* They have undergone breast surgery or breast biopsy within the last 12 months.
* They have had trauma to the breast tissue or undergone radiation treatment to the breast within the last 12 months.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female subjects who are undergoing Myocardial Perfusion imaging in the Nuclear Cardiology laboratory at the Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Biopsy-proven breast cancer | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Rhodes, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States